CLINICAL TRIAL: NCT06011395
Title: Smart Watch Insights to Prevent Exacerbations and Recurrence - Rehabilitation Study: SWIPER-REHAB
Brief Title: Smart Wearable Insights to Prevent Exacerbations and Recurrence - Rehabilitation Study: SWIPER-REHAB
Acronym: SWIPER-REHAB
Status: Not yet recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 22HH7635
Record Dates: First submitted 2023-08-21; First posted 2023-08-25 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Cardiovascular Diseases
Keywords: Cardiac rehabilitation; Prevention; Digital health; Smart wearables; Remote patient monitoring
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Smartwatch — Activity tracker (step count, calories burned), heart rate monitor
Device: Imperial Healthy Hearts app — Digital cardiac rehabilitation smartphone application. Represents smart watch data and source of educational materials for cardiac rehabilitiation programme.

SUMMARY:
Aims of the study:

* To measure the rate of completion of a digital cardiac rehabilitation programme at Imperial College Healthcare NHS Trust (ICHNT)
* To measure the health economic impact of a digital cardiac rehabilitation programme at ICHNT

Any adult patient eligible for ICHNT cardiac rehabilitation (CR) programmes is eligible to participate. Participants will receive a commercially available smart watch and be asked to wear the device as much as possible. In addition, they will be asked to download a smartphone application called 'Imperial Healthy Hearts', which displays movement and information on heart rate, breathing and oxygen levels to both the participant and the research team (digital data). The Healthy Hearts app also allows the direct care team to provide educational materials to patients as part of their routine care.

The clinical content and structure of the CR programme is determined by the clinical CR team, and does not deviate from established local and national standards and practices.

Researchers will capture physiological data such as heart rate, respiratory rate, blood pressure (where available) and oxygen saturation (where available) via the Healthy Hearts platform. Researchers will also capture clinical information from the electronic health record, and will compare CR programme uptake and completion rates with historical data and national targets.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or above
* Able to give informed consent
* Eligible for Cardiac Rehabilitation programme

Exclusion Criteria:

* Any wrist wound, skin pathology or other feature that would prohibit the wearing of a smartwatch
* Any visual impairment preventing the use of the Fitbit or smartphone application.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients at Imperial College Healthcare NHS Trust eligible for cardiac rehabilition
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2025-01-30 (Estimated); Primary Completion 2026-03-02 (Estimated); Study Completion 2026-03-02 (Estimated)

PRIMARY OUTCOMES:
Uptake of cardiac rehabilitation | 12 months
  Percentage uptake of cardiac rehabilitation programme (of those that are eligible)

SECONDARY OUTCOMES:
Quality of life assessment (EQ-5D-5L) | 12 months
  Patient quality of life as measured by the EQ-5D-5L instrument

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas S Peters, MD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided